CLINICAL TRIAL: NCT02012868
Title: Effect of Bariatric Surgery on Obstructive Sleep Apnea in a Danish Cohort
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jeppe Gram, Doctor, PhD, University of Southern Denmark
Other Study IDs: S-20120004jln
Record Dates: First submitted 2013-11-26; First posted 2013-12-16 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnoea (OSA)
Keywords: obstructive sleep apnoea; weight loss; bariatric surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Weight Loss | interventions — Bariatric Surgery; Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bariatric surgery, obstructive sleep apnoea: bariatric surgery
  Interventions: Procedure: bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgery
  Other Names: gastric bypass

SUMMARY:
Studies have shown high prevalence (60-94%) of obstructive sleep apnoea (OSA) among patients undergoing bariatric surgery.

Fifteen studies are published investigating the effect of bariatric surgery on OSA. All of them conclude a highly positive effect on OSA by bariatric surgery and weight loss. However these studies are biased by a huge number of drop outs. The drop out rate in the studies are around 60 percent.

The Investigators state that the prevalence of OSA among patients undergoing bariatric surgery in Denmark is high. The Investigators state that the effect of bariatric surgery is significant on severity of OSA. The Investigators state that we can perform a study without a huge number of dropouts.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a clinical syndrome characterized by occlusion of upper airways during sleep. The occlusions results in shortly hypoxia, which awakes the patient. When the patient awakes, activity in the pharyngeal muscles results in opening of the upper airway again.

OSA is associated with overweight. Studies have shown high prevalence (60-94%) of obstructive sleep apnea (OSA) among patients undergoing gastric bypass (bariatric) surgery.

Fifteen studies have investigated the effect of bariatric surgery on OSA. All of them conclude a highly positive effect on OSA by bariatric surgery and the following weight loss. However, a huge number of dropouts biases these studies. The dropout rate in the studies are around 60 percent. No studies are from northern Europe.

The Investigators want to perform a study investigating the prevalence of OSA among over weighted patients undergoing bariatric surgery in Denmark.

The Investigators state that the prevalence of OSA among patients undergoing bariatric surgery in Denmark is high. The investigators state that the effect of bariatric surgery is significant on severity of OSA. The Investigators state that they can perform a study without a huge number of dropouts.

The investigators investigate patients by making sleep monitoring by embletta. During one night of sleep with this apparatus, the investigators will get information on number of wake-ups during sleep, the apnea-hypopnea index and saturation during sleep. All of this gives the investigators information whether the patient have OSA or not.

Patients will undergo sleep monitoring prior to surgery. The time interval from monitoring to day of surgery varies from 1 month to one day. the investigators repeat the sleep monitoring one year after date of surgery. Differences in primary endpoint and secondary endpoints is calculated.

Today all of the subjects have undergone surgery. From November 1.2013 the investigators invites all patients to sleep monitoring once again. The investigators were hot able to register this trial before this date because of the political situation in the US. This site was closed. The Investigators hope that the investigators still are able to register the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* attending bariatric surgery

Exclusion Criteria:

* retrognathia
* micrognathia,
* acromegaly
* downs syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients attending bariatric surgery
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AHI | Change from baseline in AHI at one year
  Obstructive sleep apnoea is defined by the apnoea/hypopnoea index (AHI). This can be accessed by embletta monitoring during sleep.

SECONDARY OUTCOMES:
weight | Change from baseline in weight at one year
  No need.
Circumference of neck | Change from baseline in Circumference at neck at one year
  Circumference of the neck measured in inches.
mean saturation during sleep | Change from baseline in mean saturation during sleep at one year
  saturation during sleep is measured by a pulsoxymetry.

OTHER OUTCOMES:
ESS score | Change from baseline in ESS score at one year
  ESS is a questionnaire that gives an impression on quality of sleep. High score indicate poor quality of sleep. Low score indicate high quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lage-Hansen, Doctor, Principal Investigator — Department of endocrinology, Esbjerg
Locations (1):
- Department of endocrinology, Southern west hospital, Esbjerg, Denmark